CLINICAL TRIAL: NCT01417897
Title: Human Insulin Analogs: Evaluation of Inflammatory mRNA Expression of Macrophages and Endothelial Function of Short-acting Insulin - HERMES Pilot Study
Acronym: HERMES
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: ikfe-CRO GmbH (Industry)
Collaborators: IKFE Institute for Clinical Research and Development (Other)
Responsible Party: Principal Investigator, Marcus Borchert, Thomas Forst, MD PhD, ikfe GmbH, Clinic, ikfe-CRO GmbH
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APIDR_L_05719
Record Dates: First submitted 2011-08-15; First posted 2011-08-16 (Estimated); Last update posted 2012-03-05 (Estimated); Status verified 2012-03

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — insulin glulisine; Insulin Aspart; Insulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Insulin Glulisine: bolus injections before each main meal (Experimental): Patients are already on an Insulin Glargine therapy when they start and will them after randomization receive additionally Insulin Glulisine bolus injections before each of the main meals.
  Interventions: Drug: Insulin glulisine
- Insulin Aspart: bolus injections before each main meal (Active Comparator): Patients are already on an Insulin Glargine ± metformin therapy when they start the start and will them after randomization receive additionally Insulin Aspart bolus injections before each of the main meals.
  Interventions: Drug: Insulin aspart
- Regular human insulin:bolus injections before each main meal (Active Comparator): Patients are already on an Insulin Glargine ± metformin therapy when they start the start and will them after randomization receive additionally regular human insulin bolus injections before each of the main meals.
  Interventions: Drug: Regular human insulin

INTERVENTIONS:
Drug: Insulin glulisine — Dosage will be pro re nata. Patients should aim an blood glucose level of 2h ppBG ≤ 135 mg/dL.
  Other Names: Apidra
  Arms: Insulin Glulisine: bolus injections before each main meal
Drug: Insulin aspart — Dosage will be pro re nata. Patients should aim an blood glucose level of 2h ppBG ≤ 135 mg/dL.
  Other Names: NovoRapid
  Arms: Insulin Aspart: bolus injections before each main meal
Drug: Regular human insulin — Dosage will be pro re nata. Patients should aim an blood glucose level of 2h ppBG ≤ 135 mg/dL.
  Other Names: InsumanRapid
  Arms: Regular human insulin:bolus injections before each main meal

SUMMARY:
The planned HERMES study is to investigate and compare the effects of Insulin Glulisine, Insulin Aspart and regular human insulin on postprandial nitrotyrosine concentrations and several clinical and laboratory markers of postprandial endothelial cell function, sub-clinical inflammation and cardiovascular risk in patients with type 2 DM. The primary parameter in this study are the postprandial changes in the nitrotyrosine concentrations, a biomarker for oxidative stress. As vascular data on Insulin Glulisine vs. Insulin Aspart are missing, it is not possible to calculate sample size and statistical power. Therefore the goal of the HERMES-Pilot-Study is to generate preliminary data for statistical considerations and estimations on the probability of success of HERMES.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus
* Stable BOT (basal oral therapy) with Insulin Glargine + ≥ 2 OHA (oral hypoglycemic agents except for TZD) for a minimum of three months before entering the study
* HbA1c ≤ 8.5%
* Age between 30 and 75 years inclusively
* Body mass index ≤ 40 kg/m2
* Patient consents that his/her family physician will be informed of trial participation

Exclusion Criteria:

* Type 1 diabetes mellitus
* Unspecific infection or inflammation (hsCRP >10mg/L in POC test)
* Use of thiazolidinediones within the last 3 months prior to study start
* Retinopathy, hepatic or renal dysfunction or clinically relevant other major diseases
* History of drug or alcohol abuse within the last five years prior to screening
* History of hypersensitivity to the study drugs (or any component of the study drug) or to drugs with similar chemical structures
* History of severe or multiple allergies
* Treatment with any other investigational drug within 3 months prior to screening
* Progressive fatal disease
* hepatic (ALAT and/or ASAT > 3 times the normal reference range), renal (creatinine > 1.3 mg/dl in women and > 1.6 mg/dl in men), neurological, psychiatric and/or hematological disease as judged by the investigator
* Pregnant or lactating women
* Sexually active women of childbearing potential not consistently and correctly practicing birth control by implants, injectables, combined oral contraceptives, hormonal intrauterine devices (IUDs), sexual abstinence or vasectomized partner
* Lack of compliance or other similar reason that, according to investigator, precludes satisfactory participation in the study

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2011-09; Primary Completion 2012-05 (Estimated); Study Completion 2012-05 (Estimated)

PRIMARY OUTCOMES:
Nitrotyrosine | Baseline, after 10 weeks, after 24 weeks
  The difference in the percent increase of the oxidative stress biomarker nitrotyrosine after stimulation with a standardized meal

SECONDARY OUTCOMES:
Skin blood flow | Baseline, after 10 weeks, after 24 weeks
  Change in skin blood flow during stimulation by a standardized meal
mRNA expression of proinflammatory cytokines (MAPK/eNOS, adiponectin, hsCRP, MMP-9) | Baseline, after 10 weeks, after 24 weeks
  Biomarkers of sub-clinical inflammation and cardiovascular risk: Change in Macrophage activation, MAPK/eNOS production levels, adiponectin and hsCRP (after test meal) from baseline to endpoint
Insulin | Baseline, after 10 weeks, after 24 weeks
  Change in Insulin and the ratio from baseline to endpoint
HbA1c | Baseline, after 10 weeks, after 24 weeks
  Blood glucose control: Change during test meal, HbA1c and FBG from baseline to endpoint
Fasting blood glucose | Baseline, after 10 weeks, after 24 weeks
  Blood glucose control: Change during test meal, HbA1c and FBG from baseline to endpoint
Hypoglycemic events | Baseline, after 10 weeks, after 24 weeks
  Incidence of hypoglycemia from baseline to endpoint
intact Proinsulin | Baseline, after 10 weeks, after 24 weeks
  Change in intact Proinsulin and the ratio from baseline to endpoint

CONTACTS AND LOCATIONS:
Locations (1):
- ife GmbH, Clinic, Mainz, Rhineland-Palatinate, Germany